CLINICAL TRIAL: NCT03291158
Title: A Phase 1, Randomized, Open-Label Trial Evaluating the Plasma, Epithelial Lining Fluid, and Alveolar Macrophage Concentrations of Intravenous Minocin (Minocylcine) for Injection
Brief Title: Safety and PK Trial Evaluating the Plasma, Epithelial Lining Fluid, and Alveolar Macrophage Concentrations of Minocin IV
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Rempex Pharmaceuticals (a wholly owned subsidiary of The Medicines Company) (Industry)
Collaborators: Universitätsklinikum Köln (Other); Innovative Medicines Initiative (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDCO-MIN-16-04
Record Dates: First submitted 2017-09-18; First posted 2017-09-25 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Normal Healthy Volunteers
Keywords: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Minocycline IV (Experimental): Open label Minocin IV
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Subjects will be assigned into 5 cohorts of 5 subjects each, who will receive six doses of Minocin IV every 12 hours, starting on Day 1. Each dose of Minocin IV will be administered as an IV infusion over 1 hour. Subjects will be assigned to cohort based on time of bronchoalveolar lavage.
  Other Names: Minocin IV

SUMMARY:
This is a phase 1, safety and PK Open-Label trial evaluating the plasma, epithelial lining fluid, and alveolar macrophage concentrations of intravenous Minocin® (Minocycline) for injection in healthy adult subjects.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety of Minocin IV and measure plasma, epithelial lining fluid, and alveolar macrophage drug levels after six doses of Minocin IV given 12 hours apart, administered as 1-hour infusions in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. A signed informed consent form, the ability to understand the study conduct and tasks that are required for study participation, and a willingness to cooperate with all tasks, tests, and examinations as required by the protocol, whether in the hospital or after discharge, for the duration of the study;
2. Healthy adult male or female between 18 and 55 years of age (inclusive) at the time of Screening;
3. Body mass index (BMI) ≥ 18.5 and ≤ 30 (kg/m2) and weight between 55.0 and 100.0 kg (inclusive) at Screening;
4. Subject is in good health based on medical history and physical examination findings and has no clinically meaningful safety laboratory abnormalities (hematology, blood chemistry, and urinalysis) or 12-lead ECG results, as assessed by the Principal Investigator (PI);
5. Vital signs (blood pressure [BP], pulse, and temperature) measured at Screening/baseline must be within the following ranges: systolic BP ≥90 to ≤150 mm Hg, diastolic BP ≥45 to ≤90 mm Hg; Heart Rate ≥ 45 to ≤90 bpm (taken after resting in a supine position for at least 5 minutes);
6. Expectation that intravenous access will be sufficient to allow for ease of study drug infusion and for all protocol-required blood sampling to take place;
7. Subject commits to remaining under observation of the study staff for the course of the study;
8. Female subject is surgically sterile (bilateral tubal occlusion), postmenopausal, or if of childbearing potential, agrees to abstinence or to use a highly efficient method of birth control (i.e., intrauterine device [IUD] or intrauterine hormone-releasing system [IUS] or vasectomized male partner, or hormonal contraceptives [estrogen and progestogen combined or progestogen only] with inhibition of ovulation; oral hormonal contraceptives must be supplemented with the use of condoms), between inclusion and for 7 days after the completion of the study;
9. If male, agree to be sexually abstinent or agree to use an approved method of contraception (e.g., condom with spermicide) when engaging in sexual activity from study check-in through 7 days after completion of the study, and to not donate sperm during this same period of time.

Exclusion Criteria:

1. Has any condition, including findings in the medical history or in pre-study assessments that constitutes a risk or a contraindication for the participation in the study or completing the study;
2. Any acute illness, including clinically significant infection within 30 days prior to Day 1;
3. Surgery within the past three months prior to Day 1 determined by the PI to be clinically relevant;
4. Positive breath test for alcohol on Day 1 (pre-dose) and/or positive urine test for drugs of abuse at Screening/Day -1 visit;
5. Has a history or presence of alcohol/drug abuse within 2 years. Alcohol abuse is defined as regularly consuming >3 units/day (21 units per week for men) and >2 units/day (14 units/week) for women. A unit is defined as a can of 4% beer (330 mL), approximately 190 mL of 6-7% beer (malt liquor), a glass of 40% spirits (30 mL), or a glass of wine (100 mL);
6. Subject is a smoker and smokes >5 cigarettes per day (or equivalent);
7. Use of non-tobacco/nicotine-containing products within 6 months prior to Day 1;
8. Current diagnosis of or positive at Screening for HIV and/or Hepatitis B;
9. Blood or plasma donation within past 2 months;
10. Females who are pregnant or nursing or who have a positive pregnancy test result at Screening;
11. Presence of known raised intracranial pressure;
12. Use of isotretinoin;
13. History of significant hypersensitivity or allergic reaction to tetracycline antibiotics;
14. History of allergic or other serious adverse reactions to lidocaine;
15. Clinically significant pulmonary or any other disease that prevents a subject from undergoing bronchoscopy with bronchopulmonary lavage;
16. History of seizures (e.g., epilepsy), head injury, or meningitis requiring ongoing anti-seizure medications;
17. Receipt of any investigational medication or investigational device during the last 30 days prior to randomization;
18. Vigorous exercise from 48 hours prior to Day -1 until the day of discharge from the study;
19. Treatment with any prescription or over-the-counter drugs, within two weeks of day 1, with the exception of acetaminophen/paracetamol for minor headache. Birth control or other hormone replacement is also permitted as long as it has been taken at a stable dose for at least three months before the Screening visit and remains stable for the duration of the study;
20. Unable or unwilling to comply with the protocol;
21. An employee of the PI or study center with direct involvement in the proposed study or other studies under the direction of that PI or study center, or a family member of the employee or the PI

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Analyze plasma, ELF and Alveolar Macrophage concentrations of minocycline | 16 weeks
  Determine plasma ELF and Alveolar Macrophage concentrations of minocycline when administered to healthy adult subjects.

SECONDARY OUTCOMES:
Safety and Tolerability | 16 weeks
  To assess the safety and tolerability of Minocin IV when administered to healthy adult subjects by assessing adverse events, changes from baseline in physical examination findings, clinical safety laboratory test results, ECGs, and vital signs throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Zeitlinger, MD, Principal Investigator — University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No